CLINICAL TRIAL: NCT02237833
Title: Cerebral Oxygenation in Septic Patients Using Vasopressors - The Conscious Study
Acronym: CONSCIOUS
Status: Terminated | Type: Observational
Why Stopped: Too slow recruitment.
Sponsor: Karl-Andre Wian (Other)
Responsible Party: Sponsor-Investigator, Karl-Andre Wian, MD, Sykehuset i Vestfold HF
Organization: Sykehuset i Vestfold HF (Other)
Other Study IDs: 2014/194 REK
Record Dates: First submitted 2014-09-08; First posted 2014-09-11 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Septic Shock
Keywords: septic shock; cerebral oximetry; vasopressor; norepinephrine
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Septic shock and vasopressor: Measuring cerebral oxymetry (SCO2) first 24 hours in septic shock and given vasopressors.

SUMMARY:
The purpose of this study is to reveal if higher doses of vasopressors in septic shock patients correlates with cerebral vasoconstriction and lower cerebral oximetry.

DETAILED DESCRIPTION:
The mortality with septic shock is high. Treatment includes antibiotics, intravenous fluid and drugs for circulatory support, especially the vasopressor norepinephrine. Fluids and drugs for circulatory support are to restore adequate organ perfusion. Inadequate oxygenation of the brain can give neurologic damage. Traditionally treatment is guided by surrogate markers like arterial and central venous pressure. Cerebral oximetry is a non-invasive method which measures cerebral saturation of oxygen, SCO2, and thereby expresses regional cerebral perfusion. By registering cerebral oxymetry on patients treated with vasopressors for septic shock we want to reveal if higher doses of vasopressor correlates with cerebral vasoconstriction and lower cerebral oximetry.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Septic shock patients in ICU department requiring vasopressor therapy

Exclusion Criteria:

* Damage to the frontal lobes corresponding to the area where SCO2 is monitored
* Patients in pharmacological studies
* Patients with known intracranial vascular anomalies or cerebral aneurysms
* Patients where vasoactive medication is started before cerebral oxymetry is established
* Patients with known neurological disease
* Patients with undergone cerebral insult, transient ischemic attack or carotid stenosis
* Patients who have been resuscitated after cardiac arrest in connection with this hospital stay
* Patients with a body temperature below 35 degrees Celsius when establishing monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the intensive care unit needing vasopressor for septic shock.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of minutes of SCO2-values lower than 50 or reduced by 20% during 24 hours | 24 hours
  SCO2 will be measured before initiating vasopressor therapy. Thereafter SCO2 are updated every 2 seconds and is measured for 24 hours.

SECONDARY OUTCOMES:
Incidence of acute myocardial infarction | Hospital discharge, expected 12 days at average
  Incidence of acute myocardial infarction based on international criteria
Use of vasopressors/inotropes | Discharge from ICU, expected 5 days at average
  Use of vasopressors/inotropes
  * norepinephrine
  * epinephrine
  * dopamine
  * dobutamine
  * vasopressin
  * nitroprusside
  * glyceryltrinitrate
Fluid balance | 24 hours
Length of stay in ICU | Discharge from ICU, expected 5 days at average
Length of stay in hospital | Discharge from hospital, expected 10 days at average
Incidence of organ failure | Discharge from ICU, expected 5 days at average
  Measuring Sequential Organ Failure Assessment, SOFA, score at inclusion and once daily during ICU-stay.

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Andre Wian, cand.med., Principal Investigator — Syekhuset Vestfold HF
Locations (1):
- Sykehuset i Vestfold HF, Tønsberg, Vestfold, Norway